CLINICAL TRIAL: NCT00919841
Title: Sequential Volume Measurement of Postpartum Uterus Using 3-dimensional Sonographies
Acronym: 3DUT
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Tuangsit Wataganara, MD, Faculty of Medicine Siriraj Hospital
Other Study IDs: Si 059/2551(EC3)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: postpartum; involution; three-dimension sonography; size of the uterus
MeSH Terms: interventions — Postpartum Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postpartum women: Women who deliver a singleton vaginally
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Sequential three-dimension sonographic examination for the uterine size after vaginal delivery. The examination will be performed once a week, until the completion of 7 weeks after delivery.
  Other Names: Three dimensional ultrasound; postpartum

SUMMARY:
Women who naturally deliver a singleton will be invited to participate the study. Weekly transabdominal and/or transvaginal ultrasound examinations will be offered until the uterus is completely involuted. The pattern of involution will be analyzed.

DETAILED DESCRIPTION:
Women who naturally deliver a singleton in the Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital will be invited to participate the study. Weekly transabdominal and/or transvaginal ultrasound examinations will be offered until the uterus is completely involuted. Transabdominal or transvaginal approach will be at the examiner's discretion. Uterine volume will be measured with 3-dimensional sonographic technologies. Ovaries will also be assessed, along with Doppler flow in several vessels in the pelvis. The pattern of involution will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver a singleton vaginally will be invited to participate the study.

Exclusion Criteria:

* Women who deliver multiple gestation.
* Women who deliver by Cesarean section
* Women who have puerperal complications eg. postpartum hemorrhage or infection

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who deliver a singleton vaginally will be invited to participate the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To create the uterine involution curve after vaginal delivery | 7 weeks

SECONDARY OUTCOMES:
To assess an alteration in Doppler parameters in arcuate, uterine and ovarian arteries after vaginal delivery | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tuangsit Wataganara, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Wataganara T, Phithakwatchara N, Komoltri C, Tantisirin P, Pooliam J, Titapant V. Functional three-dimensional sonographic study of the postpartum uterus. J Matern Fetal Neonatal Med. 2015;28(18):2221-7. doi: 10.3109/14767058.2014.983063. Epub 2014 Nov 27. PMID 25363015